CLINICAL TRIAL: NCT03470441
Title: A Phase 2A, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study of Intravenous FDY-5301 in Acute Myocardial Infarction
Brief Title: A Study of Acute Myocardial Infarction Using FDY-5301
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Faraday Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: FDY-5301-201-US
Record Dates: First submitted 2018-02-27; First posted 2018-03-20 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2021-11

CONDITIONS: Acute Myocardial Infarction; STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: All subjects who fulfill all study eligibility criteria will be randomized to receive one of the 4 treatments.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blind study where all study staff and participants are blinded to whether the patient receives active drug or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- FDY-5301 Low Dose (Experimental): Anticipated n=20
  Interventions: Drug: FDY-5301
- FDY-5301 Intermediate Dose (Experimental): Anticipated n=20
  Interventions: Drug: FDY-5301
- FDY-5301 High Dose (Experimental): Anticipated n=20
  Interventions: Drug: FDY-5301
- Placebo (Placebo Comparator): Anticipated n=20
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: FDY-5301 — FDY-5301 will be administered once, intravenously, by a healthcare professional. Dosage will be administered on a body weight basis, according to treatment assignment and using the subject's body weight determined on the dose administration day.
  Arms: FDY-5301 High Dose; FDY-5301 Intermediate Dose; FDY-5301 Low Dose
Other: Placebo — Placebo will be administered intravenously by a healthcare professional. Dosage will be administered on a body weight basis, according to treatment assignment and using the subject's body weight determined on the dose administration day.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and pharmacokinetics (PK) of three dose levels of FDY-5301 compared to placebo in STEMI patients undergoing PCI.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and effectiveness of an experimental drug called FDY-5301 as a possible treatment to reduce the size of the injury to the heart caused by the heart attack. An experimental drug is one that is being tested and is not approved by the United States Food and Drug Administration (FDA).

A heart attack occurs when a heart (coronary) artery supplying blood to the heart muscle becomes blocked and the heart muscle is injured. You will be having a cardiac catheterization procedure to clear the blockage in your coronary artery that caused your heart attack. This procedure works well but may not completely prevent some injury to the heart muscle which occurs when the blood supply is initially restored to the heart. This is known as "reperfusion injury".

FDY-5301 is a single intravenous injection. About 80 subjects are expected to participate in this study at about 20 research sites in the United States and Europe. Each subject's participation is expected to last about 6 months after receiving the study drug.

Subjects who meet all inclusion criteria will be randomly assigned to one of 4 study groups. Three groups will receive FDY-5301 (low, intermediate, or high dose) and 1 group will receive a placebo.The study drug (FDY-5301 or placebo) will be given through a vein (intravenously) during the catheterization procedure. This is a double-blind study so neither the patient nor study personnel will know whether the dose is active drug or placebo until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 year old male subjects
2. 18 to 80 year old female subjects who are not of child-bearing potential.
3. Accepted for Primary PCI with diagnosis of first STEMI, based on clinical and ECG criteria (ST-elevation at the J-point in two contiguous leads with the cut-off points: ≥0.2 millivolt (mV) in men or ≥0.15 mV in women in leads V2-V3 and/or ≥0.1 mV in other leads), within 12 hours of symptom onset.

Written informed consent prior to study participation (either by the subject or a legally authorized representative of the subject)

Exclusion Criteria:

1. Previous myocardial infarction
2. Left bundle branch block (LBBB)
3. Previous coronary artery bypass graft surgery (CABG)
4. Major hemodynamic instability or uncontrolled ventricular arrhythmias
5. Known contraindication to CMR
6. Patients with known thyroid disease
7. Subjects with past or current renal impairment requiring dialysis
8. Pregnant or females of child bearing potential
9. Body weight > 120 kg or Body Mass Index (BMI) > 35 kg/m2
10. Use of investigational drugs or devices within 30 days prior to enrollment into the study.
11. Life expectancy of less than 1 year due to non-cardiac pathology
12. Any clinically significant abnormality identified at the time of screening that in the judgment of the Investigator or any sub-Investigator would preclude safe completion of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-07-14 (Actual); Study Completion 2019-01-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (2):
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Montefiore Medical Center, The Bronx, New York
- Hungary (5):
  - Budai Irgalmasrendi Kórház, Budapest
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Debreceni Egyetem Klinikai Központ, Kardiológiai és Szívsebészeti Klinika, Debrecen
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház, Miskolc
  - Zala Megyei Szent Rafael Kórház, Zalaegerszeg
- Poland (7):
  - Samodzielny Publiczny Szpital Kliniczny Nr 7 Śląskiego Uniwersytetu Medycznego w Katowicach, Górnośląskie Centrum Medyczne im. Prof. Leszka Kieca., III Oddz. Kardiologii, Katowice, Silesian Voivodeship
  - Samodzielny Publiczny Specjalistyczny Szpital Zachodnii im. Jana Pawła II, Oddział Kardiologii Inwazyjnej, Grodzisk Mazowiecki
  - Samodzielny Publiczny Specjalistyczny Szpital Zachodnii im. Jana Pawła II, Oddział Kardiologii Inwazyjnej, Krakow
  - Klinika Elektrokardiologii; Centralny Szpital Kliniczny Uniwersytetu Medycznego w Łodzi, Lodz
  - Miedziowe Centrum Zdrowia, Lubin
  - Klinika Kardiologii Inwazyjnej; Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
  - KLINIKA KARDIOLOGII, 4 Wojskowy Szpital Kliniczny, Wroclaw
- United Kingdom (9):
  - Royal Devon and Exeter Hospital Cardiology Department, Exeter, Devon
  - Wythenshawe Hospital, Manchester, Greater Manchester
  - Glenfield Hospital, Leicester, Leicestershire
  - University of Oxford, Oxford, Oxfordshire
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - New Cross Hospital, Wolverhampton, West Midlands
  - Ninewells Hospital and Medical School, Dundee
  - Royal Infirmary of Edinburgh, Edinburgh
  - Golden Jubilee National Hospital, Glasgow

REFERENCES:
- [Derived] Adlam D, Zarebinski M, Uren NG, Ptaszynski P, Oldroyd KG, Munir S, Zaman A, Contractor H, Kiss RG, Edes I, Szachniewicz J, Nagy GG, Garcia MJ, Tomcsanyi J, Irving J, Sharp ASP, Musialek P, Lupkovics G, Shirodaria C, Selvanayagam JB, Quinn P, Ng L, Roth M, Insko MA, Haber B, Hill S, Siegel L, Tulloch S, Channon KM. A Randomized, double-blind, dose ranging clinical trial of intravenous FDY-5301 in acute STEMI patients undergoing primary PCI. Int J Cardiol. 2022 Jan 15;347:1-7. doi: 10.1016/j.ijcard.2021.11.016. Epub 2021 Nov 12. PMID 34774885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant enrolled on October 27, 2017 in study centers in Poland, Hungary, UK, and the United States.
Pre-assignment Details: A total of 120 subjects were randomized 3:1 to receive one of three dosage amounts of study drug or placebo.
Groups:
- Experimental FDY-5301 Low Dose: 0.5 mg/kg FDY-5301
- Experimental FDY-5301 Intermediate Dose: 1.0 mg/kg FDY-5301
- Experimental FDY-5301 High Dose: 2.0 mg/kg FDY-5301
- Placebo: Placebo
Period: Overall Study
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Started | 29 | 31 | 31 | 29
Completed | 28 | 26 | 29 | 25
Not Completed | 1 | 5 | 2 | 4
Not completed — Death | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 4 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo | Total
Number analyzed (Participants) | 29 | 31 | 31 | 29 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 22 | 17 | 18 | 71
  >=65 years | 15 | 9 | 14 | 11 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 11 | 10 | 37
  Male | 24 | 20 | 20 | 19 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 29 | 30 | 30 | 28 | 117
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 29 | 27 | 30 | 27 | 113
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Hungary | 7 | 8 | 9 | 6 | 30
  United States | 0 | 2 | 1 | 3 | 6
  Poland | 7 | 5 | 6 | 2 | 20
  United Kingdom | 15 | 16 | 15 | 18 | 64
BMI [Mean (Standard Deviation); unit: kg/m2] | 27.1 (4.17) | 28 (4.29) | 28.1 (4.88) | 28.5 (4.43) | 27.9 (4.43)
Height [Mean (Standard Deviation); unit: cm] | 173 (7.8) | 171 (8.2) | 170 (10.7) | 170 (8.3) | 171 (8.8)
Weight [Mean (Standard Deviation); unit: kg] | 81.62 (14.703) | 81.76 (13.453) | 81.52 (15.749) | 82.23 (15.162) | 81.78 (14.601)

OUTCOME MEASURES:

1. Primary Outcome: Arrhythmias of Interest, 48 Hours (Overall)
Description: Number of patients experiencing clinically relevant arrhythmias during the first 48 hours post-treatment.
Time Frame: First 48 hours post-treatment
Measure: Number; unit: participants
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 28 | 29 | 29 | 26
participants
  Ventricular Fibrillation | 0 | 0 | 0 | 0
  Sustained Ventricular Tachycardia | 0 | 0 | 0 | 0
  Non-Sustained Ventricular Tachycardia | 1 | 1 | 7 | 2
  High-Degree AV Block | 0 | 0 | 2 | 0
  Atrial Fibrillation | 0 | 2 | 1 | 1
Statistical Analysis 1: Comparison: Experimental FDY-5301 Low Dose vs Experimental FDY-5301 Intermediate Dose vs Experimental FDY-5301 High Dose vs Placebo; Test type: Other; descriptive; As little data exists on the incidence of arrhythmias that occur over an extended period of time following AMI, descriptive analysis of the primary endpoints (Arrhythmias of Interest at 48 hours and 14 days for overall and anterior infarcts) was appropriate in this study due to the absence of an externally validated benchmark which would normally serve as the basis for hypothesis testing of FDY-5301's effect on arrhythmias

2. Primary Outcome: Arrhythmias of Interest Incidence Rate, 48 Hours (Overall)
Description: Incidence rate of clinically relevant arrhythmias during the first 48 hours post-treatment defined as the number of patients who experienced an arrhythmia divided by the total person-monitoring time within each treatment group
Time Frame: 48 hours post-treatment
Measure: Number; unit: Percentage
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 28 | 29 | 29 | 26
Percentage
  Ventricular Fibrillation | 0 | 0 | 0 | 0
  Sustained Ventricular Tachycardia | 0 | 0 | 0 | 0
  Non-Sustained Ventricular Tachycardia | .0766 | .0797 | .548 | .168
  High-Degree AV Block | 0 | 0 | .157 | 0
  Atrial Fibrillation | 0 | .159 | .0783 | .0838

3. Primary Outcome: Arrhythmias of Interest, 14 Days (Overall)
Description: Number of patients experiencing clinically relevant arrhythmias 48 hours to 14 days post-treatment.
Time Frame: 48 hours to 14 days Post Percutaneous Coronary Intervention (PCI)
Measure: Number; unit: participants
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 28 | 28 | 28 | 25
participants
  Ventricular Fibrillation | 0 | 0 | 0 | 0
  Sustained Ventricular Tachycardia | 0 | 0 | 0 | 0
  Non-Sustained Ventricular Tachycardia | 0 | 1 | 0 | 0
  High-Degree AV Block | 0 | 0 | 2 | 0
  Atrial Fibrillation | 3 | 2 | 2 | 1

4. Primary Outcome: Arrhythmias of Interest Incidence Rate, 14 Days (Overall)
Description: Incidence rate of clinically relevant arrhythmias 48 hours to 14 days post-treatment defined as the number of patients who experienced an arrhythmia divided by the total person-monitoring time within each treatment group
Time Frame: 48 hours to 14 days Post Percutaneous Coronary Intervention (PCI)
Measure: Number; unit: Percentage
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 28 | 28 | 28 | 25
Percentage
  Ventricular Fibrillation | 0 | 0 | 0 | 0
  Sustained Ventricular Tachycardia | 0 | 0 | 0 | 0
  Non-Sustained Ventricular Tachycardia | 0 | 0.0147 | 0 | 0
  High-Degree AV Block | 0 | 0 | 0.0295 | 0
  Atrial Fibrillation | 0.0475 | 0.0293 | 0.0295 | 0.0166

5. Secondary Outcome: Infarct Size Relative to Ventricular Volume, 72 Hours (Overall)
Description: Infarct size relative to ventricular volume (INF/VV) at 72 hours post-treatment
Time Frame: 72 hours post-treatment
Measure: Median (Full Range); unit: INF/VV (%)
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 22 | 18 | 20 | 20
INF/VV (%) | 19.1 [0 to 50.2] | 16.9 [0 to 51.3] | 19.6 [5.2 to 51.4] | 20.4 [0 to 60.3]

6. Secondary Outcome: Infarct Size Relative to Ventricular Volume, 3 Months (Overall)
Description: Infarct size relative to ventricular volume (INF/VV) at 3 months post-treatment)
Time Frame: 3 months post-treatment
Measure: Median (Full Range); unit: INF/VV (%)
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 24 | 14 | 22 | 15
INF/VV (%) | 11.7 [0 to 52] | 11.4 [0 to 50.7] | 8.5 [0 to 49.5] | 14.9 [0 to 48.4]
Statistical Analysis 1: Comparison: Experimental FDY-5301 Low Dose vs Experimental FDY-5301 Intermediate Dose vs Experimental FDY-5301 High Dose vs Placebo; Wilcoxon Mann-Whitney Test comparing placebo to FDY-5301 treated subjects (combined low dose, intermediate dose, and high dose); Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -3.2, 95.15% CI 2-sided [-10.8 to 3.1]

7. Secondary Outcome: Infarct Size Relative to Ventricular Volume, 72 Hours (Anterior Infarcts)
Description: Infarct size relative to ventricular volume (INF/VV) at 72 hours post-treatment)
Time Frame: 72 hours post-treatment
Measure: Median (Full Range); unit: INF/VV (%)
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 9 | 6 | 7 | 7
INF/VV (%) | 33 [0 to 39.9] | 15.8 [0 to 51.3] | 12.1 [9.8 to 45.8] | 26.7 [0 to 60.3]

8. Secondary Outcome: Infarct Size Relative to Ventricular Volume, 3 Months (Anterior Infarcts)
Description: Infarct size relative to ventricular volume (INF/VV) at 3 months post-treatment)
Time Frame: 3 months post-treatment
Measure: Median (Full Range); unit: INF/VV (%)
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 11 | 6 | 7 | 6
INF/VV (%) | 19.7 [0 to 52] | 10.4 [0 to 50.7] | 9.3 [0 to 34.4] | 22.8 [1.4 to 48.4]
Statistical Analysis 1: Comparison: Experimental FDY-5301 Low Dose vs Experimental FDY-5301 Intermediate Dose vs Experimental FDY-5301 High Dose vs Placebo; Wilcoxon Mann-Whitney Test Comparing placebo to anterior infarcts FDY-5301 treated subjects (low, intermediate, and high) combined into one group; Test type: Superiority; p = 0.46, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -4.4, 95.16% CI 2-sided [-20.2 to 12.10]

9. Secondary Outcome: Left Ventricular End Systolic Volume Index, 72 Hours (Overall)
Description: Left ventricular end systolic volume index (LVESVi) at 72 hours post-treatment
Time Frame: 72 hours post-treatment
Measure: Median (Full Range); unit: mL/kg/M2
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 25 | 21 | 21 | 21
mL/kg/M2 | 40 [20 to 65.2] | 32 [15 to 72] | 32 [12 to 68] | 38 [18 to 53]

10. Secondary Outcome: Left Ventricular End Systolic Volume Index, 3 Months (Overall)
Description: Left ventricular end systolic volume index (LVESVi) at 3 Months post-treatment
Time Frame: 3 months post-treatment
Measure: Median (Full Range); unit: mL/kg/M2
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 24 | 16 | 23 | 17
mL/kg/M2 | 29 [15 to 78] | 25.5 [7 to 100] | 27 [10 to 73] | 36 [14 to 67]

11. Secondary Outcome: Left Ventricular End Systolic Volume Index, 72 Hours (Anterior Infarcts)
Description: Left ventricular end systolic volume index (LVESVi) at 72 Hours post-treatment
Time Frame: 72 hours post-treatment
Measure: Median (Full Range); unit: mL/kg/M2
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 10 | 7 | 8 | 7
mL/kg/M2 | 45.5 [21 to 65.2] | 32 [15 to 48] | 31 [13.1 to 41] | 42 [18 to 53]

12. Secondary Outcome: Left Ventricular End Systolic Volume Index, 3 Months (Anterior Infarcts)
Description: Left ventricular end systolic volume index (LVESVi) at 3 Months post-treatment
Time Frame: 3 months post-treatment
Measure: Median (Full Range); unit: mL/kg/M2
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 11 | 6 | 8 | 7
mL/kg/M2 | 37 [16 to 68] | 28 [7 to 43] | 23.5 [14 to 40] | 36 [19 to 67]

13. Secondary Outcome: Left Ventricular Ejection Fraction, 72 Hours (Overall)
Description: Left ventricular ejection fraction at 72 hours post-treatment
Time Frame: 72 hours post-treatment
Measure: Median (Full Range); unit: Percentage
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 25 | 21 | 21 | 21
Percentage | 51.4 [31.2 to 69.5] | 51.7 [33.8 to 78.6] | 54.5 [35.9 to 75.1] | 48.7 [35.2 to 73.5]

14. Secondary Outcome: Left Ventricular Ejection Fraction, 3 Months (Overall)
Description: Left Ventricular Ejection Fraction at 3 Months (Overall)
Time Frame: 3 months post-treatment
Measure: Median (Full Range); unit: Percentage
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 24 | 16 | 23 | 17
Percentage | 59.5 [29 to 72.4] | 58.9 [25 to 87.5] | 63.2 [36.8 to 72.1] | 53.9 [39.1 to 76.9]
Statistical Analysis 1: Comparison: Experimental FDY-5301 Low Dose vs Experimental FDY-5301 Intermediate Dose vs Experimental FDY-5301 High Dose vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 3.7, 95.11% CI 2-sided [-3.6 to 10.6]

15. Secondary Outcome: Left Ventricular Ejection Fraction, 72 Hours (Anterior Infarcts)
Description: Left ventricular ejection fraction at 72 hours post-treatment
Time Frame: 72 hours post-treatment
Measure: Median (Full Range); unit: Percentage
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 10 | 7 | 8 | 7
Percentage | 48 [34.4 to 69.5] | 51.7 [33.8 to 78.6] | 57.3 [35.9 to 75.1] | 43.2 [35.2 to 73.5]

16. Secondary Outcome: Left Ventricular Ejection Fraction, 3 Months (Anterior Infarcts)
Description: Left Ventricular Ejection Fraction at 3 Months (Anterior Infarcts)
Time Frame: 3 months post-treatment
Measure: Median (Full Range); unit: Percentage
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 11 | 6 | 8 | 7
Percentage | 55.7 [34.9 to 72.4] | 57.2 [45.2 to 87.5] | 67.6 [48 to 72.1] | 50.4 [41.2 to 76.9]
Statistical Analysis 1: Comparison: Experimental FDY-5301 Low Dose vs Experimental FDY-5301 Intermediate Dose vs Experimental FDY-5301 High Dose vs Placebo; Wilcoxon Mann-Whitney Test comparing placebo to anterior infarcts FDY-5301 treated subjects (combined low dose, intermediate dose, and high dose); Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 4.9, 95.16% CI 2-sided [-7 to 16.9]

17. Secondary Outcome: Serum Troponin Concentrations, 48 Hours (Overall)
Description: Area under the curve of serum troponins measured over 48 hours post-treatment
Time Frame: 48 hours post-treatment
Measure: Median (Full Range); unit: AUC4-48 µg/L
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 25 | 25 | 24 | 19
AUC4-48 µg/L | 90.5 [-19.3 to 383] | 98.1 [0.0274 to 538] | 108 [32.8 to 591] | 112 [4.5 to 752]

18. Secondary Outcome: Serum Troponin Concentrations, 48 Hours (Anterior Infarcts)
Description: Area under the curve of serum troponins measured over 48 hours post-treatment
Time Frame: 48 hours post-treatment
Measure: Median (Full Range); unit: AUC4-48 µg/L
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 12 | 9 | 9 | 8
AUC4-48 µg/L | 123 [-19.3 to 3361] | 55 [0.0274 to 538] | 111 [32.8 to 591] | 83.8 [42.5 to 752]

19. Secondary Outcome: ST-segment Resolution
Description: Proportion of patients with ST-segment resolution at 4 hours post-dose
Time Frame: 4 hours post-dose
Measure: Number; unit: percentage
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
Number analyzed (Participants) | 25 | 25 | 21 | 19
percentage | 48.0 | 68.0 | 52.4 | 47.4

ADVERSE EVENTS:
Time Frame: Day 1 to 3 months
Arm/Group | Experimental FDY-5301 Low Dose | Experimental FDY-5301 Intermediate Dose | Experimental FDY-5301 High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 1/31 | 1/31 | 1/29
Serious Adverse Events (participants affected / at risk) | 7/29 | 7/31 | 4/31 | 8/29
Other Adverse Events (participants affected / at risk) | 9/29 | 4/31 | 9/31 | 18/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental FDY-5301 Low Dose (N=29) | Experimental FDY-5301 Intermediate Dose (N=31) | Experimental FDY-5301 High Dose (N=31) | Placebo (N=29)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery perforation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vascular stent thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental FDY-5301 Low Dose (N=29) | Experimental FDY-5301 Intermediate Dose (N=31) | Experimental FDY-5301 High Dose (N=31) | Placebo (N=29)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Haematoma (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We have multiple agreements (through our CRO) with multiple PIs in various countries. The most restrictive of those agreements prohibits the PI from publicly disclosing any study results without our (or our CRO's) prior written permission to do so.

DOCUMENTS (2):
  • Study Protocol (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT03470441/Prot_002.pdf
  • Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT03470441/SAP_003.pdf